CLINICAL TRIAL: NCT06368856
Title: Pharmacology of Mupirocin in Nasal Application in Healthy Volunteers: Monocentric Study
Acronym: MUPIPHARM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20CH024; 2020-006105-30 (EudraCT Number)
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Staphylococcus Aureus Infection
Keywords: Staphylococcus Aureus; Mupirocin; Pharmacokinetic
MeSH Terms: conditions — Staphylococcal Infections | interventions — Mupirocin

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, open-label pharmacokinetic study of mupirocin in 40 healthy subjects with 2 randomization :
  * first randomization - single dose part : 50mg or 500mg of mupirocin
  * wash-out: one month
  * second randomization - repeated doses part: 50mg mupirocin twice a day or 50 mg 3 times a day 500mg mupirocin twice a day or 500mg mupirocin 3 times a day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single dose part : 50mg mupirocin (Active Comparator): - Single dose part = single dose of 50 mg mupirocin in each nostril
  Interventions: Drug: Mupirocin (50 mg); Biological: blood samples after Single dose part; Diagnostic Test: nasal swab after Single dose part; Other: Collection of urine after Single dose part
- Single dose part : 500mg mupirocin (Experimental): Single dose part = single dose of 500 mg mupirocin in each nostril
  Interventions: Drug: Mupirocin (500 mg); Biological: blood samples after Single dose part; Diagnostic Test: nasal swab after Single dose part; Other: Collection of urine after Single dose part
- Repeated dose part: Group 1 - 50 mg of mupirocin twice a day (Experimental): 50 mg of mupirocin in each nostril twice a day (morning and evening) for 5 days
  Interventions: Drug: Mupirocin (50 mg); Diagnostic Test: nasal swab during Repeated dose part; Other: Collection of urine during Repeated dose part; Other: nasal swab after Repeated dose part
- Repeated dose part: Group 2 50 mg of mupirocin 3 times a day (Experimental): 50 mg of mupirocin in each nostril 3 times a day (morning, noon and evening) for 5 days
  Interventions: Drug: Mupirocin (50 mg); Diagnostic Test: nasal swab during Repeated dose part; Other: Collection of urine during Repeated dose part; Other: nasal swab after Repeated dose part
- Repeated dose part: Group 3 500 mg of mupirocin twice a day (Experimental): 500 mg of mupirocin in each nostril twice a day (morning and evening) for 5 days
  Interventions: Drug: Mupirocin (500 mg); Diagnostic Test: nasal swab during Repeated dose part; Other: Collection of urine during Repeated dose part; Other: nasal swab after Repeated dose part
- Repeated dose part: Group 4 500 mg of mupirocin 3 times a day (Experimental): 500 mg of mupirocin in each nostril 3 times a day (morning non and evening) for 5 days
  Interventions: Drug: Mupirocin (500 mg); Diagnostic Test: nasal swab during Repeated dose part; Other: Collection of urine during Repeated dose part; Other: nasal swab after Repeated dose part

INTERVENTIONS:
Drug: Mupirocin (50 mg) — 50 mg de mupirocin
  Other Names: Bactroban
  Arms: Repeated dose part: Group 1 - 50 mg of mupirocin twice a day; Repeated dose part: Group 2 50 mg of mupirocin 3 times a day; Single dose part : 50mg mupirocin
Drug: Mupirocin (500 mg) — 500 mg de mupirocin
  Other Names: Bactroban
  Arms: Repeated dose part: Group 3 500 mg of mupirocin twice a day; Repeated dose part: Group 4 500 mg of mupirocin 3 times a day; Single dose part : 500mg mupirocin
Biological: blood samples after Single dose part — 3 blood samples will be performed sampling time ater application of mupirocin (single dose part): 00h30, 1h00, 02h00
  Arms: Single dose part : 500mg mupirocin; Single dose part : 50mg mupirocin
Diagnostic Test: nasal swab after Single dose part — 7 nasal swab for the detection of S. aureus (type Swab) will be performed after application of mupirocin (single dose part): 00h00, 1h00, 02h00, 04h00, 06h00, 08h00, 12h00
  Other Names: intranasal concentrations
  Arms: Single dose part : 500mg mupirocin; Single dose part : 50mg mupirocin
Other: Collection of urine after Single dose part — Collection of urine during 12 hours after the application of mupirocin (Single dose part)
  Arms: Single dose part : 500mg mupirocin; Single dose part : 50mg mupirocin
Diagnostic Test: nasal swab during Repeated dose part — 5 nasal swab for the detection of S. aureus (type Swab) will be performed during administration of mupirocin (Repeated dose part): 2, 3, 4, 5 et 6 days after the first application of mupirocin (Repeated dose part)
  Arms: Repeated dose part: Group 1 - 50 mg of mupirocin twice a day; Repeated dose part: Group 2 50 mg of mupirocin 3 times a day; Repeated dose part: Group 3 500 mg of mupirocin twice a day; Repeated dose part: Group 4 500 mg of mupirocin 3 times a day
Other: Collection of urine during Repeated dose part — 5 collections of urine during Repeated dose part: 2, 3, 4, 5 et 6 days after the first application of mupirocin (Repeated dose part)
  Arms: Repeated dose part: Group 1 - 50 mg of mupirocin twice a day; Repeated dose part: Group 2 50 mg of mupirocin 3 times a day; Repeated dose part: Group 3 500 mg of mupirocin twice a day; Repeated dose part: Group 4 500 mg of mupirocin 3 times a day
Other: nasal swab after Repeated dose part — 2 nasal swab for the detection of S. aureus (type Swab) will be performed: 1, 3 months after the first application of mupirocin (Repeated dose part)
  Arms: Repeated dose part: Group 1 - 50 mg of mupirocin twice a day; Repeated dose part: Group 2 50 mg of mupirocin 3 times a day; Repeated dose part: Group 3 500 mg of mupirocin twice a day; Repeated dose part: Group 4 500 mg of mupirocin 3 times a day

SUMMARY:
Mupirocin is an old antibiotic used topically since the 1970s. Initially used in the treatment of skin infections for its antistaphylococcal action, it is now part of the decolonization strategy for Staphylococcus aureus (SA) carriage, in association with chlorhexidine. This decolonization strategy has been recommended in France for preoperative cardiac surgery in nasal SA carriers since 2013 by the French Hospital Hygiene Society, and recommended for cardiac and orthopedic surgery in SA carriers by the World Health Organization (WHO) since 2016. This strategy includes nasal decolonization using mupirocin ointment nasally (2 to 3 applications/day), a daily shower with chlorhexidine soap and + /- mouthwashes all over 5 days, often pre-operatively.

As a result, mupirocin is now widely used throughout the world, all the more so as, for reasons of ease of organization, many centers use this decolonization procedure universally (i.e. without prior screening for Staphylococcus aureus carriage), thus further increasing the use of this molecule.

Mupirocin administration methods are very vague, ranging from 2 to 3 applications per day and the application of "a match head", i.e. 50 mg, to 500 mg per nostril.

Mupirocin is bacteriostatic at low doses, becoming bactericidal at higher concentrations; low concentrations could favor the selection of resistance, so using the most effective dosage seems essential. This lack of precision in administration is linked to an almost complete ignorance of the pharmacokinetics of mupirocin and its metabolite (monic acid) after nasal application.

It therefore seems essential to conduct a pharmacokinetic study of this molecule, in order to eventually offer patients the regimen with the administration methods offering the best characteristics in terms of dosage and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject affiliated or entitled to a social security plan
* Subject having signed the consent to participate in the study

Exclusion Criteria:

* Pregnancy in progress
* Acute or chronic rhinorrhea
* Allergy to mupirocin calcium or excipients
* Any medication taken during the week preceding the beginning of the study
* Notable medical history (cardiovascular, pulmonary, neurological pathology, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
plasma concentrations of mupirocin | 0 hours 30 after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
plasma concentrations of mupirocin | 1 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
plasma concentrations of mupirocin | 2 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
intranasal concentrations of mupirocin | 1 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
intranasal concentrations of mupirocin | 2 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
intranasal concentrations of mupirocin | 4 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
intranasal concentrations of mupirocin | 6 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
intranasal concentrations of mupirocin | 8 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics
intranasal concentrations of mupirocin | 12 hours after mupirocin application (Single dose part)
  mupirocin pharmacokinetics

SECONDARY OUTCOMES:
presence of Staphylococcus aureus | Days: 5 after mupirocin application (Repeated dose part)
  Measured by nasal swab results
presence of Staphylococcus aureus | Days: 6 after mupirocin application (Repeated dose part)
  Measured by nasal swab results
presence of Staphylococcus aureus | Days: 30 after mupirocin application (Repeated dose part)
  Measured by nasal swab results
presence of Staphylococcus aureus | Days: 90 after mupirocin application (Repeated dose part)
  Measured by nasal swab results
urinary concentrations of monic acid | Days: 2 after mupirocin application (Repeated dose part)
  Analysis collection urine.
urinary concentrations of monic acid | Days: 3 after mupirocin application (Repeated dose part)
  Analysis collection urine.
urinary concentrations of monic acid | Days: 4 after mupirocin application (Repeated dose part)
  Analysis collection urine.
urinary concentrations of monic acid | Days: 5 after mupirocin application (Repeated dose part)
  Analysis collection urine.

CONTACTS AND LOCATIONS:
Overall Officials: Kasra AZARNOUSH, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No